CLINICAL TRIAL: NCT06160687
Title: Randomised Control Trial to Study the Role of Non-invasive Ventilation Using Pressure Support Ventilation Versus Adaptive Support Ventilation With Intellisync Mode in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: PSV Versus ASV With Intellisync Mode for Delivery of NIV in AECOPD
Acronym: PAINT-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM-1129
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COPD Exacerbation Acute; COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSV arm (Active Comparator): Delivery of NIV using PSV mode
  Interventions: Procedure: PSV mode during NIV
- ASV intellisync arm (Experimental): Delivery of NIV using Intelllisync ASV
  Interventions: Procedure: ASV intellisync

INTERVENTIONS:
Procedure: PSV mode during NIV — NIV will be delivered using PSV mode of ventilation
  Arms: PSV arm
Procedure: ASV intellisync — ASV intellisync mode will be used to deliver NIV
  Arms: ASV intellisync arm

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (COPD) is defined acute worsening of respiratory symptoms requiring additional therapy. COPD exacerbations affects the health status and quality of life of affected patients. The inpatient mortality during exacerbation is 3 to 4% while, intensive care unit (ICU) mortality approaches 43 to 46%. Each episode of exacerbation increases the risk of mortality subsequently(1) Non-invasive ventilation (NIV) therapy has established role in mild to moderate exacerbations of COPD. But the use of NIV therapy outside of acute exacerbation is uncertain(2) NIV use has been shown to prevent endotracheal intubation and improved hospital and ICU survival. NIV decreases the work of breathing by unloading the respiratory muscles through assisting the inspiratory phases and counterbalancing the intrinistic positive end expiratory positive pressure (ipeep)(3).

NIV is delivered through face mask, although newer interfaces like helmet available(3). Tradionally pressure targeted mode is used in NIV therapy and is often given intermittently rather than continuously(4). NIV therapy via face mask was first used by Meduri et. Al in acute respiratory failure patients. Subsequent multiple randomized control trials established the role of NIV therapy in better gas exchange, reducing PCO2, reducing endotracheal intubation thereby reducing mortality, length of stay in hospital(3).

NIV-PSV (pressure support ventilation) consists of 2 pressures. IPAP (inspiratory positive airway pressure) and EPAP (expiratory positive airway pressure) or PEEP. Pressure support is usually the pressure added above PEEP. Pressure support is usually started with 8-10 cm H2O to obtain a tidal volume of 6-8ml/kg ideal body weight. EPAP/PEEP is adjusted to counterbalance the iPEEP. It is usually kept at 4-6cm H2O. Fio2 is kept to maintain saturation of 88-92%. Inspiratory trigger is usually set at 1 L/min. Expiratory trigger kept at 50%. Back up rate should always be kept usually lower than the patient respiratory rate 10-12 breaths/min(5).

Adaptive support ventilation (ASV) is a new method of closed loop ventilation which can switch back between pressure support and pressure control modes of ventilation. Based on the ideal body weight and % of minute volume ventilation given, the ASV mode choses the best tidal volume and respiratory rate according to the patient lung mechanics by calculating expiratory time constant (RCe) through expiratory flow volume curve(6). Since closed loop system, being a completely automated system, prevent frequent adjustment by clinician and thereby increasing the time and capacity of medical staff. The first application of such closed loop system in mechanical ventilation was done by saxton in1953 in iron lung for regulation of etCO2(7). Studies published on ASV as non-invasive mode of ventilation is limited. In a feasibility study, it has been shown that ASV can be used in non-invasive mode of ventilation with similar results to PSV in COPD patients(8).

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease are periods of acute worsening during the course of illness which increase hospital admission and mortality. Intensive care unit admission and mortality are higher among elderly and those with co-morbidities(9).

Non-invasive methods of ventilation can be used in mild to moderate exacerbation of COPD. They prevent most of the complications of invasive mechanical ventilation and has also reduces mortality in acute exacerbations of COPD. In mild to moderate COPD exacerbations(pH-7.25 to 7.35), non-invasive ventilation (NIV) failure rate is found to be 15% to 20%. In severe COPD exacerbations, NIV failure rate approaches upto 52% to 62%(9).

Adaptive support ventilation (ASV) and pressure support ventilation (PSV) are among the non-invasive modes of ventilation used in COPD exacerbations.

Adaptive support ventilation:

Adaptive support ventilation is a closed loop ventilation in which it provides both pressure support and pressure controlled ventilation as per the patient needs(10). The mode was first described by Hewlett in 1977 in form of mandatory minute ventilation with adaptive pressure control(11). Later Dr. fleur T Tehrani invented this mode, which was later introduced in Galileo ventilator(11). This mode supports patient with pressure support when patient has spontaneous breath and when target ventilation is not reached it delivers pressure control breath to achieve adequate ventilation. In this mode, minute volume is controlled via Vt/RR combination based on respiratory mechanics of the patient to keep the work of breathing at minimum(10). This mode calculates the tidal volume and respiratory rate to be delivered by otis equation in its algorithm after %minute volume being set by the clinician to ensure effective ventilation at the alveolar level. The inputs provided by the clinician in this mode is %minute volume based on ideal body weight, ETS, flow trigger, maximum pressure limit(12). The mode after being initiated will deliver a series of 5 pressure limited breaths and deliver a inspiratory pressure15 cm h2o above the baseline pressure during which it calculates dynamic compliance, RCe, tidal volume and respiratory rate. These measurements are used to determine the initial targets of breath rate and tidal volume(12). After which based on respiratory rate and effort of the patient, inspiratory pressure, mandatory breath are adjusted automatically to meet the set %minute volume. ASV mode can be used as initiation, maintenance and weaning phases of mechanical ventilation and it provides full, partial or minimal ventilator support during any of these phases(12). The number of manual ventilatory adjustments are less compared to conventional mode of ventilation in ASV(13). Some randomized controlled trials performed in Non-COPD suggest shorter weaning time with ASV mode of ventilation. Shorter weaning is attributed to automated inspiratory pressure change according to patient efforts, thereby reducing ventilator patient dysynchrony and frequency of manual manipulation. In a randomized control study done by c. kirakli et. Al found out that in COPD patients ASV mode of ventilation(24 hours) has shorter weaning duration compared to pressure support mode of ventilation(72 hours) (p-value 0.041). But, this study has not found any difference in the duration of mechanical ventilation, length of stay in ICU, weaning failures when ASV and PSV mode were compared(p-value>0.05)(10) A randomized controlled trial conducted among 80 patients by Bialais et. al comparing safety, efficacy and workload of intellivent- ASV and conventional mode of ventilation (pressure assist mode and pressure support mode) found out that tidal volume delivery and spo2 were most of the time in the optimal range (6-10ml/kg IBW, spo2-92 to 96% for normal lung/ ARDS and 95-99% for brain injury) for intellivent-ASV compared to conventional mode of ventilation(p-value-0.001 and 0.005). However it was found that Pmax (maximum inspiratory pressure measured) was higher (24±5 versus 22±6) with intellivent-ASV mode than conventional ventilation(p-value-0.042). There was no significant difference between intellivent-ASV and conventional mode of ventilation in terms of time spent in optimal range of parameters like respiratory rate, PETCO2, PEEP, minute ventilation, FIO2 , RCexp. There was also no difference in length of mechanical ventilation, length of ICU stay, length of hospital stay, ICU mortality, hospital mortality and total mortality. There was comparative less need for ventilator adjustment with intellivent-ASV mode compared with conventional mode of ventilation(14).

A randomized control trial by kirakli et. Al among 229 patients found out that median mechanical ventilation duration until weaning(67{43-94} vs 92{61-165}) p-value-0.003, weaning duration(2{2-2} vs 2{2-80}hours p value-0.001) and total mechanical ventilation duration (4{2-6} days vs 4 {3-9} days, p value-0.016) were shorter in ASV group compared to pressure assist/control ventilation. Also the number of patients succeeding first attempt of extubation was higher in ASV group (p value-0.001). Weaning success and mortality were comparable between the two groups(15).

NIV-PSV:

Mechanical ventilation in its first form was used at the end of 1930s called tank ventilator. Later in 1950s during the polio epidemics, modern mechanical ventilators began to emerge. Intermittent positive pressure application via anaesthesia mask in treatment of acute respiratory illness was studied in motley and colleagues at Bellevue hospital in 1940s. The first application of NIV as CPAP via nasal mask to obstructive sleep apnea patients was done by Sullivan et. Al in 1981. Successful application of NIV via full face mask for respiratory failure in COPD patients, heart failure patients in 1989 avoided intubation. The use of NIV has increased with the introduction of ventilators with effective compensation for air leaks. NIV are most commonly used in obstructive sleep apnea, COPD and cardiac failure patients and to some extent in failed extubation. Although invasive mechanical ventilation has kept the NIV at second place, still it is used in above clinical settings(16).

In a study conducted by Hilbert et. Al, NIV-PSV was compared with standard medical treatment in COPD patients. It was found out that the days of ventilator assistance and length of ICU stay has significantly lower with NIV-PSV treated group (7±4 days vs 10±15 days, p<0.01) & (9±4 days vs 21±12 days, p <0.01) respectively. Also NIV support prevented tracheal intubation in acute exacerbation of COPD patients significantly (26% vs 71%) compared to standard medical therapy(17).

Randomized control study conducted by laurent et.al suggested that non-invasive ventilation compared to standard medical treatment for COPD exacerbation could reduce the intubation rates, length of stay in hospital(18). Another study by plant et. Al replicated the same results that early NIV therapy would reduce the number of intubation needed in mild to moderate exacerbation of COPD patients and improvement in paco2 and respiratory rate. This study suggested that NIV therapy can be effectively administered in general respiratory wards also(19).

NIV therapy was used in hypoxemic respiratory failure in post-abdominal surgery patients compared with oxygen therapy alone by jaber et. Al. NIV therapy has significantly reduced tracheal reintubation rates within 7 days following surgery (33.1% vs 45.5%, p value - 0.03) and also it provided more invasive ventilation free days compared with standard oxygen therapy(25.4 vs 23.2 days). Gas exchange was found to be similar with NIV and standard oxygen therapy in hypoxemic respiratory failure in this study. Also, the NIV group had fewer pulmonary infections compared with oxygen therapy group(20).

A randomized study by Nava et. Al conducted to study the effectiveness of NIV to prevent reintubation suggested that early institution of NIV after extubation especially in high risk patients ie) COPD, Cardiac failure, hypercapneic patients may prevent reintubation rates(4/48 vs 12/49, p-value-0.027). The delayed delivery of NIV after extubation can cause increase in mortality. So , timely delivery of NIV support can reduce mortality upto 60%. In this study NIV support was given atleast 8 hours/day after extubation(21).

Patient-ventilator asynchrony is well known in patients who are mechanically ventilated. Although there are no studies that suggest direct patient related outcome due to asynchrony, it is well known patient-ventilator asynchrony prolong the duration of mechanical ventilation(22). Although correlation with oesophageal pressure is the standard way of detecting the patient-ventilator asynchrony, a trained eye can detect most of the asynchronies using pressure-time or flow-time waveform analysis(23).Multiple studies has suggested better patient-ventilator interactions with adaptive support mode of ventilation requiring less manipulations from the clinician and also facilitating early liberation from mechanical ventilation compared to other modes of ventilation(24-26).

ELIGIBILITY:
Inclusion Criteria:

Consecutive subjects with AECOPD will be eligible for inclusion in the study if they meet all the following:

1. an acute (<7 days) sustained worsening of any of the patient's respiratory symptoms (cough, sputum quantity or character, dyspnea) beyond the normal day-to-day variation;
2. arterial blood gas analysis showing a PaCO2 >45 mm Hg with either pH between 7.25 and 7.35 or respiratory rate (18) >30 breaths/minute; and,
3. exclusion of other causes of acute breathlessness such as acute heart failure, pulmonary embolism, pneumonia, and pneumothorax.

Exclusion Criteria:

Patients with any one of the following criteria will be excluded from the current study:

1. Non-COPD acute hyper-capneic respiratory failure.
2. Hypotension (systolic blood pressure <90 mmHg).
3. Severe impairment of consciousness (Glasgow coma scale score <8).
4. Inability to clear respiratory secretions.
5. Abnormalities that preclude proper fit of the NIV interface (agitated or uncooperative patient, facial trauma or burns, facial surgery, or facial anatomical abnormality).
6. Subjects who have an artificial airway like tracheostomy tube or T-tube.
7. Patient already on home NIV therapy for chronic respiratory failure.
8. Failure to provide informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Non-invasive ventilation (NIV) failure | 28 days
  NIV failure will be defined by need for endotracheal intubation

SECONDARY OUTCOMES:
Mortality | 28 days
  Deaths due to any cause during 28 days
Time to NIV failure | 28 days
  Time from randomization to intubation
Duration of ventilation | 28 days
  Total duration of ventilation (non-invasive and invasive)
Physician and patient comfort using visual analog scale (VAS) | 28 days
  We will use VAS to measure physcian and patient's level of comfort
Asynchrony index | 28 days
  Asynchrony will be calculated manually
Complication | 28 days
  Complications attributed to NIV use

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory ICU, Department of Pulmonary Medicine, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided